CLINICAL TRIAL: NCT04271397
Title: Optimization of Tuberculosis Diagnosis and Management Using Four Immunological Biomarkers
Brief Title: Immunological Biomarkers in Tuberculosis Management
Acronym: OPTI-4TB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0757
Record Dates: First submitted 2019-12-23; First posted 2020-02-17 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis; Tuberculosis Infection
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tuberculosis (Other)
  Interventions: Other: Multiple blood samples
- Latent tuberculosis infection (Other)
  Interventions: Other: Single blood sample

INTERVENTIONS:
Other: Multiple blood samples — Patients with active tuberculosis will have 5 research-specific blood samples: V1, (baseline) immediately before initiating anti-tuberculosis treatment, then 4 samples during anti-tuberculosis treatment and follow-up, i.e. at 48 hours (V2), 15 days (V3), 2 months (V4) and 6 months (V5) after initiation of treatment. The total volume of each sample will be 20 mL for a total of 100 mL.
  Arms: Active tuberculosis
Other: Single blood sample — Patients with Latent tuberculosis infection will have a single specific sample of 14 mL.
  Arms: Latent tuberculosis infection

SUMMARY:
Tuberculosis (TB) is the leading cause of death by infectious disease in the world, responsible for 1.6 million deaths in 2017. The treatment of active TB requires at least a 6-month combined antibiotic regimen and can cause heavy side effects. As a consequence, treatment adherence is not optimal, particularly in primary care settings. Rapid and reliable monitoring of anti-TB treatment adherence and efficacy is critical to provide adequate patient care and curb relapse episodes and acquired drug resistance.

Investigators propose to evaluate the performance in terms of diagnosis accuracy and outcome prediction of four new biomarkers of active TB: 1) a double IGRA (Interferon Gamma Release Assay) including QuantiFERON-Gold Plus® and HBHA; 2) a whole blood transcriptomic analysis of mRNA (messenger Ribonucleic acid) expression of a panel of 150 genes; 3) a whole blood proteomic analysis; 4) an ex vivo immunophenotyping using flow and mass cytometry to characterize the lymphocyte populations.

ELIGIBILITY:
Inclusion Criteria:

Adult ≥ 18 year-old

* Patients having given written consent
* Patients accepting a follow up ≥ 6 months
* Proven active tuberculosis (positive direct examination and/or PCR)
* Latent tuberculosis infection assessed by positive IGRA

Exclusion Criteria:

* Malignant solid tumor
* Malignant hemopathy
* Solid organ transplantation or hematopoietic stem cell transplantation
* Immunosuppressive treatments (i.e. biologics, calcineurin inhibitors, corticosteroids)
* Auto-inflammatory disease
* Chronic liver diseases
* Chronic infection with HIV, HCV (hepatitis C virus) or HBV (hepatitis B virus)
* Antimycobacterial treatment initiated > 7 days
* Pregnancy or breastfeeding
* Refusal to participate to the study
* Persons deprived of their liberty by judicial or administrative decision
* Protected adults
* Patients not affiliated to health-care social security
* The homeless

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Concordance of the kinetics of biomarkers with the evolution of the disease | 6 months
  It is a composite outcome. Evolution of the disease is defined by clinical status, radiological computed tomography evolution and negation of the mycobacterial culture of routine respiratory samples.
  The biomarkers assessed are:
  1) a combination of IGRAs test (QuantiFERON-Gold Plus and HBHA); 2) a transcriptomic signature; 3) a protein signature; 4) a phenotypic signature (by implementing an immunomonitoring approach).

SECONDARY OUTCOMES:
Analytical characteristics of a combination of 2 IGRAs (QuantiFERON-TB Gold Plus (QFT-P) and HBHA) in the diagnosis / prognosis of tuberculosis disease. | 6 months
  Measurement of gamma interferon responses induced by different conditions of ex-vivo stimulation of the blood sample by specific Mtb peptides. This biomarker will be confronted with the evolution of the evolution of the disease as defined in the primary outcome measure.
Performance of an immunomonitoring test by mass or flow cytometry in the diagnosis / prognosis of tuberculosis by measuring the dynamics of the blood population of T lymphocytes over time. | 6 months
  Qualitative and quantitative monitoring of the different subpopulations of immune cells (CD4 + T cells, CD8 +(cluster of differentiation 8) T cells, MAIT, Th1, Th2, Th1, Tfh, Treg, naive, effector and memory cells) during anti-tuberculosis treatment will be carried out. The analytical characteristics (sensitivity, specificity, VPN and VPP) of this immunomonitoring tool will be determined by comparing the abundance of different cellular phenotypes with the evolution of the disease as defined in the primary outcome measure.
Evaluate the performance of a test based on the interpretation of a transcriptomic signature in plasma in the diagnosis / prognosis of TB. | 6 months
  A transcriptomic signature in plasma is a set of genes involved in the immune response specifically deregulated during the different stages of infection and disease progression.
  This assessment will be made from blood samples. The transcriptomic signature composed of 16 genes will be evaluated during the anti-tuberculosis treatment and confronted with the evolution of the disease as defined in the primary outcome measure.
Assess the performance of a test based on the interpretation of a protein signature in the diagnosis / prognosis of tuberculosis. | 6 months
  A protein signature is composed of cytokines and chemokines, also deregulated during the various stages of infection and progression of the disease.
  This assessment will be made from blood samples. The protein signature composed of cytokines / chemokines of interest (ie IP-10, TNF-a (tumor necrosis factor - a), IL-1(interleukin - 1), IL-18, IL-12, CCL4, IL-2, IFN-g (interferon - g),…) will be evaluated during the anti-tuberculosis treatment and confronted with the evolution of the disease as defined in the primary outcome measure.
Determine the achievement of target concentrations of rifampicin | 6 months
  To determine the achievement of target concentrations of rifampicin the pharmacokinetic profile of rifampicin will be evaluate by a combination of parameters such as the area under the curve, maximum and minimum concentration, clearance, volume of distribution, modeled from three concentration measurements at each visit. (V2, V3 and V4).
Establish the rate of metabolic self-induction of rifampicin | 6 months
  To establish the rate of metabolic self-induction of rifampicin the pharmacokinetic profile of rifampicin will be evaluate by a combination of parameters such as the area under the curve, maximum and minimum concentration, clearance, volume of distribution, modeled from three concentration measurements at each visit. (V2, V3 and V4).

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses - Hôpital de la Croix Rousse - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahuaud O, Genestet C, Hoffmann J, Dumitrescu O, Ader F. Opti-4TB: A protocol for a prospective cohort study evaluating the performance of new biomarkers for active tuberculosis outcome prediction. Front Med (Lausanne). 2022 Sep 14;9:998972. doi: 10.3389/fmed.2022.998972. eCollection 2022. PMID 36186786